CLINICAL TRIAL: NCT03018951
Title: Developing a Tool to Assess Frailty in Older Adults With a Diagnosis of Functional Mental Illness; Tool Development and Pilot Testing.
Brief Title: Assessing Frailty in Older Adults With Functional Mental Illness
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: REC REF:16 LO 1506; 196557 (Other: IRAS Project ID)
Record Dates: First submitted 2016-09-28; First posted 2017-01-12 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2019-08

CONDITIONS: Frailty; Mental Illness
Keywords: frailty, assessement
MeSH Terms: conditions — Frailty; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tool Development Stage: Older adults aged ≥65 years with a diagnosis of functional mental illness who show some signs of potentially being frail (presence of ≥2 of the following frailty indicators: Aged ≥75 years old, prescribed ≥5 medications, a history of ≥1 fall/s in the 6-month period prior to assessment, admission to hospital in the 6-month period prior to assessment. In receipt of weekly support for Activities of Daily Living (ADL) tasks, In receipt of daily support for Instrumental Activities of Daily Living (IADL) tasks, ≥2 chronic physical health conditions).
  Interventions: Other: Tool Development meeting
- Pilot Test 1: Older adults aged ≥65 years with a diagnosis of functional mental illness who show some signs of potentially being frail (presence of ≥2 of the following frailty indicators: Aged ≥75 years old, prescribed ≥5 medications, a history of ≥1 fall/s in the 6-month period prior to assessment, admission to hospital in the 6-month period prior to assessment. In receipt of weekly support for Activities of Daily Living (ADL) tasks, In receipt of daily support for Instrumental Activities of Daily Living (IADL) tasks, ≥2 chronic physical health conditions).
  Interventions: Other: Pilot Test 1 assessment session
- Pilot Test 2: Older adults aged ≥65 years with a diagnosis of functional mental illness who show some signs of potentially being frail (presence of ≥2 of the following frailty indicators: Aged ≥75 years old, prescribed ≥5 medications, a history of ≥1 fall/s in the 6-month period prior to assessment, admission to hospital in the 6-month period prior to assessment. In receipt of weekly support for Activities of Daily Living (ADL) tasks, In receipt of daily support for Instrumental Activities of Daily Living (IADL) tasks, ≥2 chronic physical health conditions).
  Interventions: Other: Pilot Test 2 assessment session

INTERVENTIONS:
Other: Tool Development meeting — Consenting participants will be invited to attend up to four meetings concerning the design of the specialist tool to assess frailty in older adults with a diagnosis of functional mental illness. The meetings will be small with up to three participants and the Chief Investigator present. The Chief Investigator will present the group with plans and ideas for the proposed assessment tool and facilitate discussions relating to these ideas. Participants will be encouraged to share their opinions and any ideas they may have. The chief investigator will take written meeting minutes during each session, which will be checked and agreed on by all meeting attendees. Each meeting will last no more than 90 minutes.
  Groups: Tool Development Stage
Other: Pilot Test 1 assessment session — Consenting participants will engage in a one off assessment session where the newly devised specialist tool to assess frailty in older adults with a diagnosis of functional mental illness will be administered. Participants will be asked a series of verbal questions related to frailty indicators and asked to engage in basic observational tests of walking speed and both static and dynamic balance. Qualitative data will be gathered from the participant to establish the comprehensibility, relevance, acceptability and feasibility of the tool via a questionnaire that includes both Likert scales and open ended questions. To assess the comprehensibility of the tool's questions each participant will also be asked to rephrase a subset of the tools questions. The duration of the assessment session will be 90 minutes maximum.
  Groups: Pilot Test 1
Other: Pilot Test 2 assessment session — Consenting participants will engage in a one off assessment session where the revised specialist tool to assess frailty in older adults with a diagnosis of functional mental illness will be administered. The administration of the tool will follow the same process as in pilot test 1. Participants will then be asked to complete a further self-rated frailty assessment tool: the Tilburg Frailty Indicator. Again, following the administration of the tools, qualitative data will be gathered from the participant to establish the comprehensibility, relevance, acceptability and feasibility of the revised tool as per the methods in pilot test 1. The tool will be scored by a study researcher and the study's chief investigator at the same time to assess inter-rater reliability. The duration of the assessment session will be 90 minutes maximum.
  Groups: Pilot Test 2

SUMMARY:
The purpose of this study is the development of, and two stages of pilot testing of, a tool designed to assess frailty in older adults with a diagnosis of a functional mental illness. During the tool's development stage, participants' input, ideas and feedback will be sought to inform the tool's design. In the first pilot test the comprehensibility, acceptability and feasibility of the tool will be established. The tool will be amended based on information gained in the first pilot test. In the second pilot test the comprehensibility, acceptability and feasibility of the revised tool will be established. Reliability of the tool will be explored and preliminary examinations of both the interpretability and construct validity of the tool will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years
* Diagnosis of one of the following functional mental illnesses; depression, anxiety, bipolar affective disorder, schizophrenia.
* Currently in receipt of mental health services under The Care Programme Approach (CPA).
* Presence of ≥2 of the following frailty indicators: Aged ≥75 years old, prescribed ≥5 medications, a history of ≥1 fall/s in the 6-month period prior to assessment, admission to hospital in the 6-month period prior to assessment. In receipt of weekly support for Activities of Daily Living (ADL) tasks, In receipt of daily support for Instrumental Activities of Daily Living (IADL) tasks, ≥2 chronic physical health conditions.
* Fluent in English language.
* Able to provide informed consent to engage in the study.
* Able to tolerate the mental and physical demands of the study

Exclusion Criteria:

* A diagnosis of a neurodegenerative condition (e.g. mild cognitive impairment or dementia), neurological condition (e.g. stroke, Parkinson's disease) or head injury (where a loss of consciousness greater than 10 minutes is reported/recorded).
* The presence of a severe sensory impairment (e.g. registered blind or deaf).
* Presence of a developmental intellectual disability.
* Current alcohol/substance abuse or dependence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Mental Health care of Older Adult community and inpatient services, South London and the Maudsley NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire | Through study completion, an average of 1 year
  The primary outcome measure for this study is a questionnaire containing both likert scales and open ended questions designed to obtain feedback from both the participant and rater regarding the comprehensibility, acceptability and feasibility of the newly devised assessment tool designed to assess frailty in older adults with a diagnosis of functional mental illness.

SECONDARY OUTCOMES:
Intraclass Correlation Coefficient and/or Cohen's Kappa (with 95% confidence intervals) | Through study completion, an average of 1 year
  The Intraclass Correlation Coefficient and/or Cohen's Kappa (with 95% confidence intervals) of the repeated measures of the revised tool designed to assess frailty in older adults with a diagnosis of functional mental illness.
The frequency of endorsement per assessment tool item | Through study completion, an average of 1 year
  The endorsement frequency for item's of the newly devised tool to assess frailty in older adult populations with a diagnosis of functional mental illness response.
Percentage of missing/incomplete items | Through study completion, an average of 1 year
  The percentage of missing/incomplete items of the newly devised tool to assess frailty in older adult populations with a diagnosis of functional mental illness.
Correlation coefficient | Through study completion, an average of 1 year
  Correlation coefficients between scores of the revised tool designed to assess frailty in older adult with a diagnosis of functional mental illness tool and the Tilburg Frailty Indicator

CONTACTS AND LOCATIONS:
Overall Officials: Robert Howard, Professor MD, Principal Investigator — King's College London
Locations (1):
- South London and the Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sutton JL, Gould RL, Daley S, Coulson MC, Ward EV, Butler AM, Nunn SP, Howard RJ. Psychometric properties of multicomponent tools designed to assess frailty in older adults: A systematic review. BMC Geriatr. 2016 Feb 29;16:55. doi: 10.1186/s12877-016-0225-2. PMID 26927924
- [Background] Sutton JL, Gould RL, Coulson MC, Ward EV, Butler AM, Smith M, Lavelle G, Rosa A, Langridge M, Howard RJ. Multicomponent Frailty Assessment Tools for Older People with Psychiatric Disorders: A Systematic Review. J Am Geriatr Soc. 2019 May;67(5):1085-1095. doi: 10.1111/jgs.15710. Epub 2018 Dec 27. PMID 30589075